CLINICAL TRIAL: NCT00469378
Title: An Open-label Study of Leukocyte Counts in the Cerebrospinal Fluid and Blood of Subjects With Relapsing Forms of Multiple Sclerosis Following Treatment With Firategrast
Brief Title: Study Of White Blood Cells In The Cerebrospinal Fluid And Blood Of Patients With Relapsing Forms Of Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4M108119
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: firategrast; lymphocytes; leukocytes; SB-683699; cerebrospinal fluid; relapsing forms of multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Firategrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- firategrast (Experimental): 900 (females) or 1200 (males) mg twice daily for 24 weeks
  Interventions: Drug: firategrast

INTERVENTIONS:
Drug: firategrast — 900 (females) or 1200 (males) mg twice daily for 24 weeks

SUMMARY:
This is a study to count the number of white blood cells in the cerebrospinal fluid and blood at the beginning and end of treatment with firategrast and at 4 and 12 weeks after stopping firategrast. Cerebrospinal fluid flows through and protects the brain and spinal cord. It is important to understand what happens to the number of white blood cells because they are important in preventing infections.

ELIGIBILITY:
Inclusion criteria:

Specific information regarding warnings, precautions, contraindications, adverse events (AEs), and other pertinent information on the investigational product that may impact subject eligibility is provided can be found in the SB-683699 Investigators Brochure [GlaxoSmithKline Document Number HM2002/00094/05].

Subjects eligible for enrollment in the study must meet all of the following criteria:

* Written informed consent.
* Male or female, age 18 to 65.
* A diagnosis of a relapsing form of MS [As per McDonald, 2001; Polman, 2005], with dissemination in time and space.
* Expanded Disability Status Scale (EDSS) score of between 0 and 6.5 inclusive.
* Occurrence of at least one clinical attack in the previous 24 months, but not within the 4 weeks prior to Screening or prior to the Baseline Visit.
* A minimum of two T2 lesions on brain MRI at Screening, as determined by the central MRI analysis reader.
* A female subject is eligible to enter the study if she is:

  1. Of non-childbearing potential, i.e. a woman who:

     * has documented evidence of tubal ligation, bilateral oophorectomy or hysterectomy; or
     * is post-menopausal, defined as at least one year without menses in the absence of hormone replacement therapy. In questionable cases, menopausal status will be confirmed by estradiol and Follicle Stimulating Hormone (FSH) levels consistent with menopause according to local laboratory ranges. Estrogen-containing hormone replacement therapies (HRT) are not allowed during the study.

     OR
  2. Of childbearing potential, has a negative urine pregnancy test at Screening and Baseline, and agrees to consistent and correct use the method of contraception listed below. Subjects will use effective contraceptive methods for at least one month prior to Screening and should continue to use the same contraceptive method throughout the study until 3 days after the last dose of firategrast.

     * Progesterone-only oral contraceptives or implants (inserted at least one month prior to Screening, but not beyond the third successive year following insertion). Estrogen-containing contraceptives are not allowed during the study.
     * Intrauterine Device (IUD) (inserted by a qualified clinician, with published data showing that the highest expected failure rate is less than 1% per year).
     * Spermicide in conjunction with either a diaphragm, cervical cap or condom.
     * Male partner sterilization (vasectomy) prior to female subject's entry into the study and is the sole partner for that female subject.

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Subjects receiving corticosteroids within 4 weeks of Screening for treatment of MS. If non-systemic steroids are being used for other chronic inflammatory conditions, subjects may be included at the discretion of the investigator after discussion with the GSK medical monitor.
* Use of a b-interferon product, glatiramer acetate or azathioprine within 3 months of Screening, or use of Mitoxantrone within 12 months of Screening. Subjects who have received other therapies affecting the immune system (such as intravenous immunoglobulin (IVIg), cyclophosphamide, plasmapheresis, or any other immunosuppressive or immunomodulatory treatment) in the past may be included on a case by case basis after discussion with the GSK medical monitor. None of these treatments will be allowed during this study.
* Previous exposure to alemtuzumab, natalizumab or firategrast administration, bone marrow transplantation or whole body irradiation.
* Subjects with a cardiac pacemaker or any other type of metal implant or with any other contraindication for MRI (including known allergy to gadolinium).
* Use of 4-aminopyridine, rosiglitazone, pioglitazone or any drug that is an inhibitor of or a substrate (with a low therapeutic index) for Organic Anion Transporter Protein (OATP).
* Subjects with clinically significant renal laboratory values: subjects with a calculated creatinine clearance <60ml/min (by Cockcroft and Gault) at Screening [Cockcroft, 1976].
* Subjects with local urinalysis findings of 1) proteinuria, defined as ³1+ protein on urine dipstick or 2) renal tubular cell casts or 3) ³5 red blood cells / high power field will be excluded from the study if the result is still present on a repeat urinalysis during the Screening Phase.
* Presence of clinically significant hepatic laboratory values: Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Gamma Glutamyl Transferase (GGT) > 2 times the upper limit of the reference range; total bilirubin > 1.5 the upper limit of the normal range.
* CD4 count < 500, CD4:CD8 < 1.0, JCV viremia in plasma or white cells, idiopathic CD4/CD8 lymphopenia or secondary lymphopenia at Screening.
* Any findings at Screening on the MRI of the brain other than MS, except for benign findings that (in the opinion of the central MRI reading site and local site investigator) require no further evaluation or treatment and do not impact patient's neurological health (e.g. small arachnoid cysts, venous angiomas).
* Uncontrolled or any active bacterial, viral, or fungal infection. Any previous serious infections should be discussed with the GSK medical monitor (e.g. opportunistic or atypical infections).
* History of tuberculosis (TB) or positive chest X-ray for TB at Screening (prior chest X-ray is acceptable if performed within previous 6 months).
* Known congenital or acquired immunodeficiency.
* Current or history of cancer, excluding localized non-melanoma skin cancer.
* Any abnormality on 12-lead Electrocardiogram (ECG) at Screening which is clinically significant in the opinion of the investigator.
* Positive hepatitis B surface antigen, hepatitis C antibody or HIV tests at Screening.
* Women who are lactating, pregnant (positive pregnancy test at Screening), or planning to become pregnant during the course of the study.
* Recent history or suspicion of current drug abuse (including analgesic abuse) or alcohol abuse within the last 6 months prior to Screening. Alcohol abuse is defined as an average weekly intake of greater than 21 units for men and 14 units for women or an average daily intake of greater than three units for men and two units for women. One unit is equivalent to approximately 250mL of beer or one measure of spirits or one glass of wine.
* Use of an investigational drug for a condition other than MS within 30 days or 5 half-lives (whichever is longer) preceding Screening. Prior use of an investigational drug for MS should be discussed with the GSK medical monitor.
* Any concurrent illness, disability or clinically significant abnormality (including laboratory tests) that may affect the interpretation of clinical efficacy or safety data or prevent the subject from safely completing the assessments required by the protocol.
* Contraindications, in the opinion of the investigator, to lumbar puncture, e.g. congenital or acquired spine or CNS conditions that may render LPs unsafe, platelet count of less than 50 GI/L and/or an International Normalized Ratio (INR) of greater than or equal to 1.5 (by history), known history of clotting/bleeding disorder, needle phobia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Assessment of total leukocytes in cerebrospinal fluid (CSF) | Baseline (Week 0), Week 24, 28 and 36
  Total leukocyte count in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. CSF sample data presented are results from the local clinical laboratory.
Change from Baseline in number of total leukocytes in CSF | Baseline (Week 0) and Week 24, 28 and 36
  Total leukocyte count in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. CSF sample data presented are results from the local clinical laboratory. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of total leukocytes in blood | Baseline (Week 0), Week 4, 24, 28 and 36
  Total leukocyte count in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. Blood sample data presented are results from the independent assessor.
Change from Baseline in number of total leukocytes in blood | Baseline (Week 0) and Week 4, 24, 28, 36
  Total leukocyte count in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. Blood sample data presented are results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of total lymphocytes in CSF | Baseline (Week 0), Week 24, 28 and 36
  Total lymphocyte count in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor.
Change from Baseline in number of total lymphocytes in CSF | Baseline (Week 0) and Week 24, 28, 36
  Total lymphocyte count in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of total lymphocytes in blood | Baseline (Week 0), Week 4, 24, 28 and 36
  Total lymphocyte count in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor.
Change from Baseline in number of total lymphocytes in blood | Baseline (Week 0) and Week 4, 24, 28, 36
  Total lymphocyte count in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of lymphocyte subsets in CSF (CD3+CD4+CD8+, CD19+, CD3-CD16+CD56+, CD3+CD4-CD8-) | Baseline (Week 0), Week 24, 28 and 36
  The count for lymphocyte subsets CD3+CD4+CD8+ "double positives" (T-lymphocyte), CD3+CD4-CD8- "double negatives" (T-lymphocyte), CD19+ (B-lymphocyte) and CD3-CD16+CD56+ (natural killer cells) in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor.
Change from Baseline in number of lymphocyte subsets in CSF (CD3+CD4+CD8+, CD19+, CD3-CD16+CD56+, CD3+CD4-CD8-) | Baseline (Week 0) and Week 24, 28, 36
  The count for lymphocyte subsets CD3+CD4+CD8+ "double positives" (T-lymphocyte), CD3+CD4-CD8- "double negatives" (T-lymphocyte), CD19+ (B-lymphocyte) and CD3-CD16+CD56+ (natural killer cells) in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of lymphocyte subsets in blood (CD3+CD4+CD8+, CD19+, CD3-CD16+CD56+, CD3+CD4-CD8-) | Baseline (Week 0), Week 4, 24, 28 and 36
  The count for lymphocyte subsets CD3+CD4+CD8+ "double positives" (T-lymphocyte), CD3+CD4-CD8- "double negatives" (T-lymphocyte), CD19+ (B-lymphocyte) and CD3-CD16+CD56+ (natural killer cells) in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor.
Change from Baseline in number of lymphocyte subsets in blood (CD3+CD4+CD8+, CD19+, CD3-CD16+CD56+, CD3+CD4-CD8-) | Baseline (Week 0) and Week 4, 24, 28, 36
  The count for lymphocyte subsets CD3+CD4+CD8+ "double positives" (T-lymphocyte), CD3+CD4-CD8- "double negatives" (T-lymphocyte), CD19+ (B-lymphocyte) and CD3-CD16+CD56+ (natural killer cells) in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All the data presented are based on results from independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of lymphocyte subset CD4 count in CSF | Baseline (Week 0), Week 24, 28 and 36
  The count for CD4 cells in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor.
Change from Baseline in lymphocyte subset CD4 count in CSF | Baseline (Week 0) and Week 24, 28, 36
  The count for CD4 cells in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of lymphocyte subset CD4 count in blood | Baseline (Week 0), Week 4, 24, 28 and 36
  The count for CD4 cells in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor.
Change from Baseline in lymphocyte subset CD4 count in blood | Baseline (Week 0) and Week 4, 24, 28, 36
  The count for CD4 cells in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of lymphocyte subset CD8 count in CSF | Baseline (Week 0), Week 24, 28 and 36
  The count for CD8 cells in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor.
Change from Baseline in lymphocyte subset CD8 count in CSF | Baseline (Week 0) and Week 24, 28, 36
  The count for CD8 cells in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of lymphocyte subset CD8 count in blood | Baseline (Week 0), Week 4, 24, 28 and 36
  The count for CD8 cells in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor.
Change from Baseline in lymphocyte subset CD8 count in blood | Baseline (Week 0) and Week 4, 24, 28, 36
  The count for CD8 cells in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of CD4:CD8 ratio in CSF | Baseline (Week 0), Week 24, 28 and 36
  The count for CD4:CD8 ratio in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor.
Change from Baseline in CD4:CD8 ratio in CSF | Baseline (Week 0) and Week 24, 28, 36
  The count for CD4:CD8 ratio in the CSF was done at Baseline (Week 0), Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Assessment of CD4:CD8 ratio in blood | Baseline (Week 0), Week 4, 24, 28 and 36
  The count for CD4:CD8 ratio in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor.
Change from Baseline in CD4:CD8 ratio in blood | Baseline (Week 0) and Week 4, 24, 28, 36
  The count for CD4:CD8 ratio in the blood was done at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. All data presented are based on results from the independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.

SECONDARY OUTCOMES:
Assessment of CD34+ cells in the blood | Baseline (Week 0), Week 4, 24, 28 and 36
  Blood sample was examined to test the mobilization of CD34+ early hematopoietic progenitor cells from the bone marrow at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. CD34+ was measured using two different approaches by the independent assessor: a. Without a CD45 side scatter histogram (SSH) added and this analysis was conducted by the individual flow cytometry laboratories and the independent assessor and b. With a CD45 SSH added and the analysis was conducted by the independent assessor only. All the data presented are based on results from independent assessor.
Change from Baseline in number of CD34+ cells in the blood | Baseline (Week 0) and Week 4, 24, 28, 36
  Blood sample was examined to test the mobilization of CD34+ early hematopoietic progenitor cells from the bone marrow at Baseline (Week 0), Week 4, Week 24, Week 28 and Week 36. CD34+ was measured using two different approaches by the independent assessor: a. Without a CD45 SSH added and this analysis was conducted by the individual flow cytometry laboratories and the independent assessor and b. With a CD45 SSH added and the analysis was conducted by the independent assessor only. All the data presented are based on results from independent assessor. Baseline was defined at Week 0. Change from Baseline is the value at indicated time points minus the Baseline value.
Number of participants with adverse events (AEs) and Serious adverse events (SAEs) | Up to Week 24
  AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was any untoward medical occurrence that, at any dose results in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or was considered as medically significant. On-treatment AEs and SAEs have been presented.
Cumulative number of new gadolinium-enhancing lesions at Week 24 | Week 24
  The number of new gadolinium-enhancing lesions was determined by magnetic resonance imaging (MRI) scan. The cumulative number of new gadolinium-enhancing lesions at 24 weeks of treatment was derived as the sum of new gadolinium-enhancing lesions counted at all visits from Week 4 up to Week 24. In the event that a participant had missing MRI data for a gadolinium enhanced lesion parameter during the on-treatment period (scans at Weeks 4-24 inclusive), the missing value was imputed using the mean value for that parameter for all non-missing scans during the treatment period.
Cumulative volume of new gadolinium-enhancing lesions at Week 24 | Week 24
  The volume of new gadolinium-enhancing lesions was determined by MRI scan. The cumulative volume of new gadolinium-enhancing lesions was calculated at each visit from Week 4 up to Week 24. In the event that a participant had missing MRI data for a gadolinium enhanced lesion parameter during the on-treatment period (scans at Weeks 4-24 inclusive), the missing value was imputed using the mean value for that parameter for all non-missing scans during the treatment period.
Cumulative number of persistent gadolinium-enhancing lesions at Week 24 | Week 24
  The number of persistent gadolinium-enhancing lesions was determined by MRI scan. The cumulative number of persistent gadolinium-enhancing lesions at 24 weeks of treatment was derived as the sum of persistent gadolinium-enhancing lesions counted at all visits from Week 4 up to Week 24. In the event that a participant had missing MRI data for a gadolinium enhanced lesion parameter during the on-treatment period (scans at Weeks 4-24 inclusive), the missing value was imputed using the mean value for that parameter for all non-missing scans during the treatment period.
Cumulative total number of enhancing Lesions at Week 24 | Week 24
  The total number of gadolinium-enhancing lesions was determined by MRI scan. The cumulative total number gadolinium-enhancing lesions at 24 weeks of treatment was derived as the sum of the new and persistent gadolinium-enhancing lesions counted at all visits from Week 4 up to Week 24. In the event that a participant had missing MRI data for a gadolinium enhanced lesion parameter during the on-treatment period (scans at Weeks 4-24 inclusive), the missing value was imputed using the mean value for that parameter for all non-missing scans during the treatment period.
Plasma and CSF levels of firategrast | Week 24, 28 and 36
  Pharmacokinetic sampling for plasma and CSF levels of firategrast was done on Week 24 of treatment period and Week 28 and 36 of core follow up period, however the results for these parameters were not analyzed.
The relationship between plasma concentration of firategrast and lymphocyte count in the CSF | Week 24, 28 and 36
  Sampling to determine concentration of firategrast and lymphocyte count in the CSF was supposed to be done on Week 24 of treatment phase and Week 28 and 36 of core follow up period to investigate any relationship between lymphocyte counts and systemic exposure to firategrast and its metabolite GW786375X. There was no quantifiable concentrations of firategast or its metabolite GW786375X, hence, the results were not analyzed.
The relationship between plasma concentration of firategrast and lymphocyte count in the blood | Week 24, 28 and 36
  Sampling to determine concentration of firategrast and lymphocyte count in the blood was supposed to be done on Week 24 of treatment phase and Week 28 and 36 of core follow up period to investigate any relationship between lymphocyte counts and systemic exposure to firategrast and its metabolite GW786375X, however, the results were not analyzed.
The relationship between the presence of the A allele of rs887829 and bilirubin levels | Baseline (Week 0)
  Participants were assessed for the presence of A allele of rs887829 which is associated with Gilbert's syndrome. Gilbert's syndrome is benign and characterized by transient increases in bilirubin levels (>1.5XUpper limit of normal [ULN]). Participants who were carrying two copies of A allele of rs887829, suggested that elevations in bilirubin (maximum total bilirubin [MTB] >1.5xULN, >1.0 to 1.5xULN and less than or equal to 1.0xULN) were due to benign Gilbert's syndrome. Genotypes AA, AG and GG were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- GSK Investigational Site, Brussels, Belgium
- Czechia (2):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- Denmark (2):
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Koebenhavn Ø
- GSK Investigational Site, Lørenskog, Norway
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå